CLINICAL TRIAL: NCT07347002
Title: A Test-Negative Case-control Study to Evaluate the Effectiveness of VLA1553 Against Chikungunya Virus Disease During a Pilot Vaccination Strategy in Brazil
Brief Title: Observational Study to Assess the Effectiveness of VLA1553 Vaccine in Preventing Chikungunya During a Pilot Vaccination Strategy in Brazil
Status: Enrolling by invitation | Type: Observational
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: Fundação Butantan (Unknown); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Other Study IDs: VLA1553-402
Record Dates: First submitted 2025-12-04; First posted 2026-01-16 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Test-positive for Chikungunya virus
  Interventions: Biological: Live-attenuated CHIKV vaccine VLA1553
- Controls: Test-negative for Chikungunya virus
  Interventions: Biological: Live-attenuated CHIKV vaccine VLA1553

INTERVENTIONS:
Biological: Live-attenuated CHIKV vaccine VLA1553 — Non-interventional study: VLA1553 is used in the pilot vaccination strategy which is linked to this observational study.

SUMMARY:
This is an observational, non-interventional, test-negative case-control (TNCC) study to estimate the vaccine effectiveness of VLA1553 against Chikungunya virus in a real-world setting.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of vaccination with VLA1553 in the prevention of laboratory-confirmed symptomatic cases of CHIK after a single dose of VLA1553 administered as part of a pilot vaccination strategy following licensure in Brazil.

The study will commence following the implementation of the pilot vaccination strategy in selected municipalities. Data for the analyses will be obtained from official Brazilian Ministry of Health surveillance systems, specifically the GAL (Laboratory Environment Management System), SINAN (Notifiable Diseases Information System), and Si-PNI (National Immunization Program Information System).

ELIGIBILITY:
Inclusion Criteria:

1. Have place of residence in a municipality where the pilot vaccination strategy is implemented;
2. Are in an eligible age-group to receive the VLA1553 vaccine;
3. Have been notified in SINAN as a suspected case for CHIK or Dengue surveillance during the study period;
4. Have a sample registered in GAL that is collected within 0-5 days following the onset of CHIKV-like symptoms and is tested for CHIKV using RT-PCR;
5. Have complete data in the Brazilian MoH databases (SINAN and GAL) on age, sex, municipality of residence, sample collection date, and date of symptom onset and the healthcare facilities where the suspected case was reported.

Exclusion Criteria:

1. Have inconclusive RT-PCR result for CHIKV;
2. Have the first CHIKV-like symptom onset less than 14 days from date of vaccination.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Residents of the selected areas, within the age limits approved for the PVS, presenting at the health care facilities during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Detection of CHIKV in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated study individuals with CHIKV-like symptoms confirmed by reverse transcriptase polymerase chain reaction (RT-PCR). | Study start through study completion, an average of 23 months

SECONDARY OUTCOMES:
Detection of CHIKV in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated study individuals ≥50 years of age with CHIKV-like symptoms confirmed by RT-PCR. | Study start through study completion, an average of 23 months

OTHER OUTCOMES:
Detection of CHIKV in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated individuals with CHIKV-like symptoms confirmed by RT-PCR, stratified by sex and age group (≥18 to 59 and ≥ 60 years, depending on the age group approved for the PVS) | Study start through study completion, an average of 23 months
Detection of CHIKV in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated study individuals with CHIKV-like symptoms confirmed by RT-PCR, stratified by time since vaccination (from 0 to 6 months after Day 15) | Study start through study completion, an average of 23 months
CHIKV hospitalizations (confirmed by RT-PCR) in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated study individuals; CHIKV deaths (confirmed by RT-PCR) in VLA1553-vaccinated (≥14 days after vaccination) and unvaccinated study individuals | Study start through study completion, an average of 23 months
Magnitude and direction of estimated level of bias due to unmeasured pre-vaccination strategy CHIKV infection, and estimated VE corrected for this bias. | Study start through study completion, an average of 23 months

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Universidade Federal Do Ceará, Fortaleza, Ceará
  - Universidade Federal de Minas Gerais, CT Terapias Avançadas e Inovadoras, Belo Horizonte, Minas Gerais
  - Centro de Pesquisas Clínicas Universidade Federal Sergipe, Hospital e Maternidade São João de Deus, Laranjeiras, Sergipe
  - Fundação Faculdade Regional De Medicina De São José Do Rio Preto, São Pedro, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided